CLINICAL TRIAL: NCT01686282
Title: Daily Incorporation of Blueberries Into a Diet Favorably Improves Vascular Function and Lowers Aortic Blood Pressure in Postmenopausal Women With Pre- and Stage 1-hypertension.
Brief Title: Blueberry Consumption Improves Vascular Function and Lowers Blood Pressure in Postmenopausal Women With Pre- and Stage 1-hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, Bahram Arjmandi, Margaret A. Sitton Professor and Director of the Center for Advancing Exercise and Nutrition Research on Aging, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 021259
Record Dates: First submitted 2012-09-11; First posted 2012-09-18 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Arterial Stiffness; Blueberry Supplementation; Aortic Blood Pressure; Hypertension; Postmenopausal; Pulse Wave Velocity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 8 weeks of freeze-dried blueberry powder taken in two doses of 22g each per day.
  Interventions: Dietary Supplement: Placebo
- Blueberry (Experimental): 8 weeks of freeze-dried blueberry powder taken in two doses of 22g each per day.
  Interventions: Dietary Supplement: Freeze-dried Blueberry Powder

INTERVENTIONS:
Dietary Supplement: Freeze-dried Blueberry Powder — 8 weeks of freeze-dried taken in two doses of 22g each per day.
  Other Names: U.S. Highbush Blueberry Council
  Arms: Blueberry
Dietary Supplement: Placebo — 8 weeks of freeze-dried taken in two doses of 22g each per day.
  Arms: Placebo

SUMMARY:
Cardiovascular disease (CVD) continues to be the leading cause of death in the U.S. Americans have been more concerned about their blood cholesterol levels and dietary cholesterol intakes rather than their overall cardiovascular health risk factors leading to CVD such as hypertension, vascular dysfunction, inadequate consumption of fruits and vegetables and physical activity. Statistics show that approximately 91% of individuals with CVD have vascular dysfunction which is attributed to endothelial and autonomic dysfunction leading to increased arterial stiffness.

The investigators long-term goal is to provide feasible and effective dietary ways for pre- and stage 1- hypertensive individuals to normalize their blood pressure (BP), improve vascular function and thereby reducing their cardiovascular risk and enhancing the quality of life. Blueberries are a rich source of phenolic compounds and these compounds may play an important role in promoting cardiovascular health. Considering the strong possibility that phytochemicals present in blueberry work additively or synergistically, it would be ideal to investigate the cardioprotective effects of blueberry as a whole. The investigators overall objective to bring forth evidence that blueberry consumption will reduce BP and cardiovascular risk factors including endothelial dysfunction, arterial stiffness, and autonomic dysfunction in pre- and stage 1-hypertensive postmenopausal women. The investigators hypothesize that blueberry supplementation will improve vascular function and will lower blood pressure in postmenopausal women with pre-hypertension. The findings of this study will provide a foundation for disseminating feasible, safe approaches for preventing and combating hypertension at its early stage which does not require drug therapy.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of 22 grams of freeze-dried blueberry intake on a daily basis for eight weeks in:

The purpose of the study is to examine the effects of 22 grams of freeze-dried blueberry intake on a daily basis for eight weeks on arterial function and blood pressure in postmenopausal women with pre- and stage 1-hypertension. The specific aims of the study are:

1. To investigate the extent to which daily consumption of 22 g blueberry drink-mix reduces blood pressure in individuals with pre- and stage 1-hypertension.
2. To determine whether daily consumption of 22 g blueberry drink-mix will improve the autonomic control of blood pressure and heart rate in individuals with pre- and stage 1-hypertension.
3. To measure serum markers of oxidative stress to determine whether increased antioxidant defense is in part responsible for blueberry's vascular protective effects.

ELIGIBILITY:
Inclusion Criteria:

* 40 women (1 to 10 years after natural menopause or bilateral oophorectomy) 45-65 years of age.
* Seated blood pressure ≥ 130/85 mm Hg but ≤ 160/90 mm Hg.

Exclusion Criteria:

* Blood pressure >160/100 mmHg
* Taking insulin
* Cardiovascular disease
* Active cancer
* Asthma
* Glaucoma
* Thyroid disease
* Kidney disease
* Liver disease
* Pancreatic disease
* Enrollment in a weight loss program
* Heavy smokers (>20 cigarettes per day)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 8 weeks
  By measuring aortic blood pressure at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).

SECONDARY OUTCOMES:
Autonomic Control of Blood Pressure | 8 weeks
  By measuring blood pressure variability and baroreflex sensitivity at rest and during physiological stress.
Autonomic Control of Heart Rate | 8 weeks
  By measuring heart rate variability at rest and during physiological stress.
Endothelial Function | 8 week
  By measuring markers of vascular inflammation (adiponectin, leptin, endothelin-1, angiotensin II and 8-isoprostane).
Inflammation | 8 weeks
  By measuring a marker of inflammation (tumor necrosis factor-α [TNF-α]).
Oxidative Stress | 8 weeks
  By measuring markers of oxidative stress (superoxide dismutase [SOD], nitrate/nitrite [NOx], ET-1, angiotensin II, 8-isoprostane, MDA, and oxidized LDL).
Arterial Stiffness | 8 Week
  By measuring the augmentation index and arterial stiffness at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).

CONTACTS AND LOCATIONS:
Overall Officials: Bahram H Arjmandi, PhD, RD, Principal Investigator — Florida State University; Arturo Figueroa, MD, PhD, Principal Investigator — Florida State University; Sarah A Johnson, PhD, RD, CSO, Principal Investigator — Florida State University
Locations (1):
- The Department of Nutrition, Food, and Exercise Sciences, Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Johnson SA, Figueroa A, Navaei N, Wong A, Kalfon R, Ormsbee LT, Feresin RG, Elam ML, Hooshmand S, Payton ME, Arjmandi BH. Daily blueberry consumption improves blood pressure and arterial stiffness in postmenopausal women with pre- and stage 1-hypertension: a randomized, double-blind, placebo-controlled clinical trial. J Acad Nutr Diet. 2015 Mar;115(3):369-377. doi: 10.1016/j.jand.2014.11.001. Epub 2015 Jan 8. PMID 25578927